CLINICAL TRIAL: NCT07006857
Title: Comparative Effects of Exercise Combined With Music at Varying Frequencies on Physical and Cognitive Performance in Young Adults
Brief Title: Effects of Exercise With Different Music Frequencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Physical Inactivity
Keywords: Exercise; Cognition; Music Therapy; Yoga; Performance
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise with Low Frequency (Experimental)
  Interventions: Other: Low Frequency
- Exercise with High Frequency (Experimental)
  Interventions: Other: High Frequency Music
- Exercise without Music (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise without music
  Arms: Exercise without Music
Other: Low Frequency — 396 Hertz (Hz), 417 Hz, 528 Hz, 639 Hz
  Arms: Exercise with Low Frequency
Other: High Frequency Music — 741 Hz, 852 Hz, 963 Hz
  Arms: Exercise with High Frequency

SUMMARY:
This study will explore the impact of different music frequencies applied during yoga based exercises on physical performance and cognitive status in inactive young adults.

DETAILED DESCRIPTION:
This study will explore the impact of different music frequencies applied during yoga based exercises on physical performance and cognitive status in inactive young adults aged between 18-35 years. Thirty participants will be randomly assigned into three groups: low-medium frequency music, high frequency music, and a control group without music.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy woman or man between the ages of 18-35 years,
* Not having any ongoing musculoskeletal problems that prevent doing exercise/physical activity (Will be assessed with the Physical ActivityReadiness Questionnaire).
* Being physically inactive according to the International Physical Activity Short Form
* Being a volunteer to participate in the study.
* Being able to read and understand Turkish.

Exclusion Criteria:

* Ongoing pregnancy,
* Having any hearing problems or colorblindness,
* Using regular medications with potential neurological side effects (psychiatric medications, painkillers, etc.).
* Continuing treatment due to a psychiatric diagnosis such as clinical depression, anxiety, bipolar disorder, or schizophrenia.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Stroop Test | 8 weeks
  The Stroop Test is a psychological assessment that measures cognitive flexibility and processing speed by requiring individuals to name the color of the ink used for words that represent different colors, which can create interference. Lower test completion duration indicate better cognitive flexibility.

SECONDARY OUTCOMES:
Sit To Stand Test | 8 weeks
  The Sit to Stand Test is a physical assessment that evaluates lower body strength and balance by measuring how many times a person can stand up from a seated position and sit back down in a set time period. Higher repetions indicate better body strength.
Wall Squat test | 8 weeks
  The Wall Squat Test measures lower body endurance by assessing how long an individual can maintain a squat position against a wall with their back for a specified duration. Higher duration for test completation indicate good body endurance.
Push Up Test | 8 weeks
  The Push Up Test evaluates upper body strength and endurance by counting the maximum number of push-ups a person can perform in a set time or until exhaustion. Higher numbers show better strength and endurance.
Handgrip Electronic Dynamometer | 8 weeks
  The Handgrip Electronic Dynamometer measures grip strength by quantifying the force exerted when a person squeezes a handheld device, providing an objective assessment of hand and forearm strength. In scoring, higher kilograms that assessed indicate better strength.
Sit And Reach | 8 weeks
  Sit And Reach measures flexibility and hamstring length by determining how far a person can reach toward their toes while sitting with legs extended. the reached distance is assessed with measuring tape in centimeter. Exceeding toes is showed in positive values and not reaching toes is showed in negative values. Reaching far away from the foot toes indicate better flexibility, and scored with positive values.
Nelson Ruler Test | 8 weeks
  The Nelson Ruler Test evaluates hand-eye coordination and fine motor skills by having individuals use a ruler to catch it as it falls, measuring their reaction time and accuracy. Lower catching time indicate higher reaction skill.
Global Scale of Change | 8th week
  The Global Scale of Change is a tool used to measure individual perceptions of change in various contexts, often assessing the extent of improvement or deterioration in health, function, or well-being over time.

CONTACTS AND LOCATIONS:
Overall Officials: Begüm Kara Kaya, PhD, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Zeytinburnu, Istanbul, Turkey (Türkiye)